CLINICAL TRIAL: NCT03613883
Title: The Endovascular Management of Visceral Artery Aneurysms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud K. khairallah, Principal Investigator, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: endovascular in aneurysms
Record Dates: First submitted 2018-06-29; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Visceral Artery Aneurysm
Keywords: aneurysm; embolization; stent graft
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Study Arm (Experimental): The intervention is done to those patients that are managed by endovascular stent that is inserted in the parent artery to induce slowness in the blood flow thus initiate thrombosis in the aneurysmal sac.
  Interventions: Procedure: Endovascular management
- Expanded Selection Arm (Experimental): The intervention is done to the expanded selection arm and is managed by embolic materials (coils / glue) that occlude the aneurysm by proximal occlusion, proximal and distal occlusion or sac packing
  Interventions: Procedure: Endovascular management

INTERVENTIONS:
Procedure: Endovascular management — Embolic materials (coils / glue): the glue will be routinely used when access into the aneurysm's outflow vessel will be unattainable.
  Endovascular stent to slow the flow inducing thrombosis of the sac of aneurysm. CT angiography will be performed later to evaluate and confirm the diagnosis and viability of the endovascular procedure

SUMMARY:
To describe the safety, possible complications and technical success of different technical methods and different embolic materials in the endovascular management of visceral artery aneurysms.

DETAILED DESCRIPTION:
Abdominal visceral artery aneurysms (VAAs) are defined as aneurysms which involve branches of the celiac, superior mesenteric, inferior mesenteric or renal arteries. Owing to the improvements in imaging technology and the use of cross-sectional imaging modalities (ultrasound, computed tomography [CT], and magnetic resonance imaging), there is increase in the frequency of VAAs diagnosis. Although classically treated by open surgery, modern treatment strategies generally place interventional radiology techniques at the top of the treatment algorithm. Therefore, vascular interventional radiologists must become familiar with the indications for the treatment of VAA, become experienced in the different techniques, and know when to recommend treatment of VAA by interventional radiology techniques or to advocate open surgical repair.

VAAs are subdivided into true and false aneurysms. A true aneurysm involves all three layers of the arterial wall. Classically, a true aneurysm is defined as a localized dilatation of the artery by more than 1.5 times the expected arterial diameter. True aneurysms occur as a result of underlying arterial pathology such as atherosclerosis, fibromuscular dysplasia, and arteritis. The prevalence of true VAAs is 0.1-2%, and most true VAAs are asymptomatic. A minority may cause abdominal pain, which may be a harbinger of imminent rupture. VAAs are almost never large enough to be palpable by examination. False aneurysms, or pseudoaneurysms, are effectively contained ruptures of the artery that are lined by adventitia or by the perivascular tissues. False aneurysms may occur as a result of inflammation, infection, or trauma.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysm due to inflammation or pancreatitis [e.g., splenic, gastroduodenal (GDA), superiomesenteric artery (SMA), hepatic, or even renal aneurysms].
* Aneurysm due to trauma.
* Aneurysms occurring after surgery
* Aneurysm due to penetrating peptic ulcers.

Exclusion Criteria:

* In most cases with multiple, diffuse, small aneurysms related to portal hypertension should be left untreated and followed by repeat computed tomography (CT) or magnetic resonance imaging (MRI) examinations. Once the portal hypertension and underlying cirrhotic disease is treated (e.g., via liver transplantation), the aneurysm may spontaneously decrease and completely disappear over time.
* Patient refusal.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Complete aneurysm exclusion at the final angiographic control with absence of contrast extravasation and cessation of haemorrhage. | At immediate post-procedure
  Complete aneurysm exclusion at the final angiographic control with absence of contrast extravasation and cessation of haemorrhage, if originally present. In instances of aneurysmal disease of second-order or third-order branches, technical success is further defined as exclusion of the aneurysm with preservation of flow within the intended parent artery.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa H Othman, M.D., Study Director — Radiology Department in Assiut University Hospital